CLINICAL TRIAL: NCT07033507
Title: Diagnostic Performance of Combining Apparent Diffusion Coefficient and Micro-calcifications to Kaiser Score in Evaluation of BI-RADS 4 Breast Lesions
Brief Title: Diffusion Coefficient and Micro-calcifications to Kaiser Score in Evaluation of BI-RADS 4 Breast Lesions
Status: Recruiting | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abd Elmoniem Mohamed, Lecturer faculty of medicine, Mansoura University Hospital
Other Study IDs: MD.24.04.846
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Breast Neoplasms
Keywords: BI-RADS 4 breast lesions; diffusion coefficient; micro-calcifications; Kaiser Score
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BI-RADS 4 breast lesions: evaluate the reliability of ADC and micro calcifications (when present) in combination with the Kaiser score in improving the accuracy of the evaluation of BI- RADS 4 lesions and helping avoidance of unnecessary biopsies.
  Interventions: Diagnostic Test: MRI diffusion coefficient and micro-calcifications to Kaiser Score in evaluation of BI-RADS 4 breast lesions

INTERVENTIONS:
Diagnostic Test: MRI diffusion coefficient and micro-calcifications to Kaiser Score in evaluation of BI-RADS 4 breast lesions — Compare MRI diffusion coefficient and micro-calcifications to Kaiser Score in evaluation of BI-RADS 4 breast lesions

SUMMARY:
Breast cancer is the most commonly diagnosed cancer worldwide and is the leading cause of cancer-related deaths in women. Mammography, breast ultrasonography (US), and breast magnetic resonance imaging (MRI) are essential for the diagnosis and follow-up of breast cancer. The American College of Radiology Breast Imaging- Reporting and Data System (ACR BI-RADS), which is used worldwide, provides the standard terminology for breast imaging (Jajodia et al., 2021). The ACR BI- RADS lexicon categorizes breast imaging findings into seven BIRADS categories of 0, 1, 2, 3, 4(4a, 4b, 4c), 5, and 6 according to the probability of malignancy. Breast imaging findings assigned as BI-RADS 4 require tissue sampling and histopathological examination. However, the likelihood of malignancy of lesions classified as BI-RADS 4 ranges widely, from 3% to 94%. Categorization of lesions according to BI-RADS is related to the experience of the radiologist, with experienced radiologists performing better than inexperienced radiologists

DETAILED DESCRIPTION:
A method with lower inter-reader variability for distinguishing benign lesions from BI-RADS 4 lesions needs to be developed to help avoiding unnecessary biopsies. The Kaiser score (KS) is a classification tree flowchart based on machine learning, which can guide clinical decision-making about breast imaging findings on breast MRI. It selects five morphological features and kinetics among 17 categorical diagnostic criteria to score each breast lesion and applies to both mass and non-mass enhancement (NME) lesions. The KS value ranges from 1 to 11, with increasing values indicating higher probability of malignancy. A biopsy is recommended, if the lesion score exceeds 4.

Ductal carcinoma in situ (DCIS), whose incidence has recently increased rapidly, only manifests as suspicious microcalcifications from time to time. Between 70% and 90% of DCIS diagnoses depend mainly on detecting microcalcifications on mammography.The morphology and distribution of microcalcifications are of great significance in distinguishing between benign and malignant micro calcifications. Given its confinement to the milk ducts, DCIS always presents as NME lesions and may be false-negative on MRI. A previous study suggested that the KS should be upgraded in the presence of suspicious mammographic microcalcifications to avoid missed DCIS diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Patients with BI-RADS 4 lesion.

Exclusion Criteria:

* Patients on chemotherapy or related treatment.
* Patients who have contraindications to do MRI as patients with cardiac pace maker, patients with cochlear implant and ocular foreign body, claustrophobia.

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Evaluation of BI-RADS 4 breast lesions
Study Population: All patients will give age, Menstrual status and hormonal contraceptive use. Past and family history of breast cancer.
  Local breast and Axillary lymph nodes examination Imaging: MRI will be performed for BIRADS 4 lesions. Mammography will be performed for assessment of the presence of microcalcifications. Measurement of ADC value. Using the Kaiser score to re-evaluate BI-RADS 4 lesions, combined microcalcifications with Kaiser Score, combined ADC with Kaiser score.
  Mammography protocol: cranio-caudal and medio-lateral oblique. MRI protocol: using a 1.5 T magnet using a breast coil and will be done between 7th -14th days of the menstrual cycle.
  Dynamic post-contrast study Axial T1-fast spin echo Axial T2-fast spin echo Axial and coronal T2-inversion recovery
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of combining apparent diffusion coefficient and micro-calcifications to Kaiser Score in evaluation of BI-RADS 4 breast lesions | 12 months
  evaluate the reliability of ADC and micro calcifications (when present) in combination with the Kaiser score in improving the accuracy of the evaluation of BI- RADS 4 lesions and helping avoidance of unnecessary biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmoniem, Principal Investigator — Lecturer of faculty of medicine Mansoura university
Locations (1):
- Mohamed AbdElmoniem, Al Mansurah, Egypt